CLINICAL TRIAL: NCT04084405
Title: Effect of Inspiratory Muscle Training on Balance During PR in Chronic Obstructive Pulmonary Disease Patients (COPD)
Brief Title: Effect of Inspiratory Muscle Training During Pulmonary Rehabilitation on Balance in COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Medicine, Sousse (Other)
Responsible Party: Principal Investigator, Bilel Tounsi, PhD student, Faculty of Medicine, Sousse
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: COPD-Balance
Record Dates: First submitted 2019-09-05; First posted 2019-09-10 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; IMT; ABC; BBS; TUG; SLS
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMT group (Experimental): Inspiratory muscle training + aerobic exercice
  Interventions: Other: Pulmonary rehabilitation
- Control group (Active Comparator): aerobic exercice
  Interventions: Other: Pulmonary rehabilitation

INTERVENTIONS:
Other: Pulmonary rehabilitation — The experimental group receives inspiratory muscle training and aerobic exercise. The Active Comparator group received only aerobic exercise.

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a respiratory disease that results in progressive airflow limitation and respiratory distress. Physiopathological features of COPD suggest that people who suffer from this disease have many risk factors for falls that have been identified in older individuals.

The benefit of inspiratory muscle training (IMT) combined with a pulmonary rehabilitation programme (PRP) is uncertain. The investigators aimed to demonstrate that,in chronic obstructive pulmonary disease (COPD) patients, IMT performed during a PRP is associated with an improvement of Balance.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease COPD is a preventable and treatable disease(GOLD, 2017). According to the WHO, COPD would be the third leading cause of death by 2030 (WHO, 2017). This disease is characterized by airflow limitation that is not fully reversible. The airflow limitation is usually progressive and associated with an abnormal inflammatory response of the lung to noxious particles or gases(GOLD, 2017). However, emerging data showed that COPD patients demonstrate important deficits in balance and control which associated to a high risk of fall ( Butcher et al, 2004 ; Smith et al, 2009 ; Beauchamp et al, 2009 ; Beauchamp et al, 2010). Inspiratory muscle training (IMT) has been shown to be an effective modality for COPD patients for improving the maximal inspiratory muscle strength, the dyspnea and health-related quality of life (GI COPD, 2016). However, the effect of inspiratory muscle training on balance is not studying. The purpose of this study is to evaluate the effect of the inspiratory muscles training on balance in COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Were COPD diagnosed by pulmonary function testing
* clinically stable
* abscence of other obstructive diseases
* signed written consert.

Exclusion Criteria:

* Were previous pneumonectomy or lobectomy in the past 6 months
* spontaneous risk of pneumothorax or rib fracture
* incapacity to follow a standard rehabilitation programme (locomotor deficits, acute cardiac failure and acute exacerbation of COPD at the beginning of the programme)
* the absence of written informed consent.

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Inspiratory muscle strengh | Baseline, 2 months follow up
  The inspiratory muscle strengh were measured by pre and post maximal inspiratory preasure
ACTIVITIES-SPECIFIC BALANCE CONFIDENCE test (ABC) | Baseline, 2 months follow up
  The ABC scale requires patients to indicate their confidence in performing 16 activities without losing their balance or becoming unsteady on an 11-point scale (0%-100%).Higher scores indicates higher balance confidence and lower scores indicates poor balance confidence
Berg Balance Scale (BBS) | Baseline, 2 months follow up
  The patients were evaluated by The test BBS. The score obtained from 0 to 56.Higher scores indicate better balance.
Single Leg Stance (SLS) | Baseline, 2 months follow up
  Patients selected the leg on which they they preferred to stand for the test. They were instructed to keep their legs from touching and to maintain a unipedal stance for as long as possible
Timed Up and Go (TUG) | Baseline, 2 months follow up
  The test requires the patient to rise from a standard armchair, walk 3 m at a comfortable pace, walk back to the chair, and sit down

SECONDARY OUTCOMES:
The six minutes walk test (6MWT) | Baseline, 2 months follow up
  The test provides estimate endurance and funcional performance of patients

CONTACTS AND LOCATIONS:
Locations (1):
- Bilel TOUNSI, Sousse, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crisan AF, Oancea C, Timar B, Fira-Mladinescu O, Tudorache V. Balance impairment in patients with COPD. PLoS One. 2015 Mar 13;10(3):e0120573. doi: 10.1371/journal.pone.0120573. eCollection 2015. PMID 25768731
- [Derived] Tounsi B, Acheche A, Lelard T, Tabka Z, Trabelsi Y, Ahmaidi S. Effects of specific inspiratory muscle training combined with whole-body endurance training program on balance in COPD patients: Randomized controlled trial. PLoS One. 2021 Sep 23;16(9):e0257595. doi: 10.1371/journal.pone.0257595. eCollection 2021. PMID 34555068